CLINICAL TRIAL: NCT05999084
Title: Georgia Memory Net Center for Medicare and Medicaid Services Registry for Anti-Amyloid Monoclonal Antibody Coverage with Evidence Development
Brief Title: Georgia Memory Net Anti-Amyloid Monoclonal Antibody Registry
Status: Recruiting | Type: Observational
Sponsor: Emory University (Other)
Collaborators: Centers for Medicare and Medicaid Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, James Lah, Associate Professor, Emory University
Other Study IDs: STUDY00006475
Record Dates: First submitted 2023-08-13; First posted 2023-08-21 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Alzheimer Disease
Keywords: Monoclonal antibodies; Amyloid; Mild Cognitive Impairment; Lecanemab; Leqembi
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — lecanemab; Standard of Care

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Anti-amyloid Monoclonal Antibodies (mAbs): Patients with Mild Cognitive Impairment (MCI) or mild AD dementia who are receiving treatment with anti-amyloid mAbs, per standard of care. Patients seen in the Emory and GMN MACs are evaluated with standard instruments for cognitive and functional abilities.
  Interventions: Drug: Anti-amyloid Monoclonal Antibodies (mAbs)
- Historical Comparator Group: Available historical data from biomarker-confirmed patients with MCI or mild dementia due to AD who have been followed in the Emory Cognitive Neurology Clinic will serve as a comparator group. Patients seen in the Emory and GMN MACs are evaluated with standard instruments for cognitive and functional abilities.
  Interventions: Combination Product: Standard of Care
- Caregivers of Patients Receiving Anti-amyloid Monoclonal Antibodies (mAbs): Caregivers of patients with Mild Cognitive Impairment (MCI) or mild AD dementia who are receiving treatment with anti-amyloid mAbs, per standard of care. Caregivers of patients seen in the Emory and GMN MACs are evaluated with standard instruments for cognitive and functional abilities.
  Interventions: Drug: Anti-amyloid Monoclonal Antibodies (mAbs)

INTERVENTIONS:
Drug: Anti-amyloid Monoclonal Antibodies (mAbs) — Infusions of lecanemab occur every 2-weeks as indicated in the FDA labeling. After 18 months of treatment, an amyloid positron emission tomography (PET) scan with FDA-approved radiotracer is performed to confirm clearance of amyloid pathology. It is anticipated that most individuals treated with lecanemab for 18 months will no longer have positive amyloid PET scans. In those instances where persistent amyloid pathology is seen, every 2-week treatment with lecanemab will be continued for an additional 6 months with repeat amyloid PET scan until amyloid clearance is achieved. If an individual has progressed to moderate or severe stages of AD dementia during the initial 18 months of treatment and amyloid PET shows failure to clear amyloid pathology, treatment will be terminated. Dosing frequency after 18 months (or after amyloid clearance) remains unclear and will need to be determined with additional evidence development.
  Other Names: lecanemab
  Groups: Anti-amyloid Monoclonal Antibodies (mAbs); Caregivers of Patients Receiving Anti-amyloid Monoclonal Antibodies (mAbs)
Combination Product: Standard of Care — The standard of care, other than treatment with anti-amyloid mAbs, provided at the study clinics.
  Groups: Historical Comparator Group

SUMMARY:
The purpose of this registry is to compile information on patients who are receiving FDA-approved anti-amyloid mAbs in the course of their clinic visits in the Emory Cognitive Neurology Clinic and in Georgia Memory Net Memory Assessment Clinics.

DETAILED DESCRIPTION:
Alzheimer's disease is a devastating neurodegenerative illness impacting millions of Americans including patients and caregivers. Treatments have been limited to symptomatic therapies leading to the pervasive sentiment that 'nothing can be done'; however, recent advances in the field have created excitement and hope for patients, families, and healthcare providers. On 6 January 2023, the anti-amyloid monoclonal antibody (mAb) lecanemab received accelerated approval from the Food and Drug Administration (FDA). A similar medication, donanemab, also recently demonstrated positive results in a large trial. Despite the positive trials, questions remain about anti-amyloid mAbs efficacy as well as how they will perform in a real-world setting. The Centers for Medicare & Medicaid Services (CMS) released a National Coverage Analysis (NCA) Memo with a framework for deploying anti-amyloid mAbs in a way that improves understanding of benefit and harm.

This registry will be managed through Georgia Memory Net (GMN), an initiative that was launched in 2018 to build statewide capacity for early and specific diagnosis of Alzheimer's disease and related dementias (ADRD), improve patient and caregiver support, and provide access to emerging disease modifying therapies. The GMN supports Memory Assessment Clinics (MACs) geographically distributed at 7 sites around the state with common data elements modeled on best practices developed in the Emory University Cognitive Neurology Memory Assessment Clinic over the past 25 years. The GMN infrastructure and care model provides an optimal real-world testing ground for evidence development on the effectiveness, safety, and appropriate use of anti-amyloid mAbs in the Medicare population.

The clinical data for patients treated with anti-amyloid mAbs will be compared to historical clinical data from comparable patients who were seen in GMN clinics prior to availability of anti-amyloid mAbs. Patients in the registry will be followed for the duration of their initial treatment as specified by FDA for specific anti-amyloid monoclonal antibody and subsequent maintenance treatment which is currently unspecified.

The objectives of this registry are to:

1. Monitor clinical use of FDA approved anti-amyloid mAbs to report health outcomes for patients in broad community practice.
2. Understand how patient characteristics, treating clinicians, and clinical settings impact benefits and harms (brain hemorrhage and edema) of FDA approved anti-amyloid mAbs.
3. Define how benefits and harms of FDA approved anti-amyloid mAbs change over time.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50-90, inclusive
2. Diagnosis: Mild Cognitive Impairment (MCI) or mild AD dementia with positive cerebrospinal fluid (CSF) or amyloid PET
3. Objective measurement of baseline cognition and function within past 3 months:

   * Cognitive: Mini-Mental State Examination (MMSE) ≥ 22, MoCA ≥ 16
   * Function: Independence in basic ADLs
   * Function: FAQ ≤ 9 may justify inclusion with lower cognitive score if felt to be impacted by prominent language impairment or other factors affecting score
4. MRI brain within last year and no exclusionary criteria
5. Complete blood count (CBC), comprehensive metabolic panel (CMP), B12, thyroid stimulating hormone (TSH), prothrombin time (PT), partial thromboplastin time (PTT), and International Normalized Ratio (INR) without clinically significant abnormality
6. Informant/care partner/family available to attend follow-up visits to provide information regarding patient's cognitive and functional abilities
7. Agree to MRI, PET, and testing clinical diagnostic requirements and drug label / FDA recommendations to determine drug eligibility and appropriateness, including Apolipoprotein E (APOE) testing

Exclusion Criteria:

1. Any contraindication to MRI
2. MRI exclusion criteria:

   * Acute or sub-acute hemorrhage
   * Prior macro hemorrhage (>1 cm), subarachnoid hemorrhage, or known aneurysm
   * >4 microhemorrhages
   * Superficial siderosis
   * Any finding that might be a contributing cause of the subject's dementia that could pose a risk to the subject or prevent safety MRIs.
3. Seizure within the past 6 months or history of refractory epilepsy.
4. Unstable severe psychiatric illness in past 6 months
5. History of bleeding disorder, blood clotting, or clinically significant abnormal results on coagulation profile (platelet count <50,000; INR >1.5)
6. Uncontrolled diabetes (HgbA1c >9%)
7. Uncontrolled hypertension
8. History of unstable angina, myocardial infarction (MI), advanced heart failure, or clinically significant conduction abnormalities within past year.
9. End stage renal disease
10. Receiving active treatment for cancer (e.g., chemotherapy, biologics, or radiation therapy) with exceptions for maintenance therapies for cancer in remission (e.g., anti-estrogen for breast cancer)
11. Systemic illness or serious infection, e.g., pneumonia, sepsis, Coronavirus disease 2029 (COVID-19), in past 30 days
12. Immunological disease requiring immunosuppression, immunoglobulins, monoclonal antibodies, or plasmapheresis
13. Exclude if breastfeeding or if female patients of childbearing potential unable to practice highly effective contraception
14. History of severe allergic or anaphylactic reactions or hypersensitivity to inactive ingredients (arginine hydrochloride, histidine, histidine hydrochloride monohydrate, polysorbate 80)

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study includes patients receiving care through the Emory Cognitive Neurology Clinic and Georgia Memory Net (GMN) clinics, and their caregivers.
Sampling Method: Non-Probability Sample
Enrollment: 735 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Change in Quick Dementia Rating System (QDRS) Score | Baseline and every 6 months until end of study (up to 5 years)
  The QDRS is a 10-item questionnaire assessing cognitive impairment. Items are rated on a 5-point scale where no problems = 0, slight problems = 0.5, mild problems = 1, moderate to severe problems = 2, and severe problems = 3. Total scores range from 0 to 30 and higher scores indicate increased cognitive impairment.
Montreal Cognitive Assessment (MoCA) Score | Baseline and every 6 months until end of study (up to 5 years)
  MoCA is an instrument to screen for mild cognitive dysfunction, assessing the cognitive domains of attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. Total scores range from 0 to 30 with higher scores indicating better cognitive function. A normal score is considered to be 26 or higher.
Change in Functional Activities Questionnaire (FAQ) Score | Baseline and every 6 months until end of study (up to 5 years)
  Instrumental activities of daily living are assessed with the Functional Activities Questionnaire (FAQ). The FAQ includes 10 items which are scored on a scale from 0 to 3 where 0 = normal and 3 = dependent. Total scores range from 0 to 30 and lower scores indicate that the respondent is able to perform daily activities. A score of 9 (where the person is dependent in 3 activities) is used as a cut-point indicating impairments with functioning.
Change in Lawton-Brody Activities of Daily Living (ADL) Physical Self-Maintenance Scale (PSMS) Score | Baseline and every 6 months until end of study (up to 5 years)
  Independence with tasks such as toilet behaviors, feeding, and grooming is measured with the Physical Self-Maintenance Scale (PSMS). The PSMS is a 6-item instrument with multiple options for responses, which are scored as 0 or 1. Complete independence with the activity is scored as 1 and if any sort of assistance is needed the score is 0 . Total scores range from 0 to 6 with higher scores indicating greater independence with tasks of self-maintenance.
Change in Lawton-Brody Instrumental Activities of Daily Living (IADL) Scale Score | Baseline and every 6 months until end of study (up to 5 years)
  Functional independence is measured with the Instrumental Activities of Daily Living (IADL) scale. The IADL is an 8-item instrument which assesses how well the respondent can perform daily tasks of using the telephone, shopping, food preparation, housekeeping, laundry, transport, medication, and finances by rating the responses as 0 or 1. The total score for women ranges from 0 to 8 and the total score for men ranges from 0 to 5, with higher scores indicating greater independence.

SECONDARY OUTCOMES:
Change in Care Needs Assessment Tool (CNAT) Score | Baseline and every 6 months until end of study (up to 5 years)
  The CNAT asks caregivers to indicate whether or not certain challenging behaviors (9 items) or difficulties with activities of daily living (4 items) have occurred with the care recipient in the past month. For the behaviors and difficulties that have happened, caregivers rate how much they were bothered by this on a 5-point scale where "not at all" = 0 and "extremely" = 4. Total score for this section range from 0 to 52, with higher scores indicating a increased feelings of being upset about the behaviors and functional difficulties of the care recipient.
Change in Zarit Burden Interview Score | Baseline and every 6 months until end of study (up to 5 years)
  The Zarit Burden Interview instrument assesses caregiver burden and needs. The measurement has 22 items about feelings while caring for another person and each item on the interview is a statement which the caregiver is asked how often they feel that way. Responses are given on a 5-point scale where Never - 0 and Nearly Always = 4. Total scores range from 0 to 88 and higher scores indicate greater feelings of burden.
Change in Patient-Reported Outcomes Measurement Information System Global Health (PROMIS 10) Score | Baseline and every 6 months until end of study (up to 5 years)
  The PROMIS Global Health questionnaire consists of 10 items assessing general domains of health and functioning. Items are scored on a 5-point scale where poor = 1 and excellent = 5. Total scores are standardized to a T-score with a mean of 50 and a standard deviation of 10. Scores above 50 indicate better health and functioning, while scores below 50 indicate physical, mental and social health that is below average.

CONTACTS AND LOCATIONS:
Overall Officials: James J Lah, MD, PhD, Principal Investigator — Emory University
Locations (8):
- United States (8):
  - Georgia Memory Net Memory Assessment Clinic - Albany, Albany, Georgia
  - Georgia Memory Net Memory Assessment Clinic - Atlanta, Atlanta, Georgia
  - Emory Clinic, Atlanta, Georgia
  - Georgia Memory Net Memory Assessment Clinic - Augusta, Augusta, Georgia
  - Georgia Memory Net Memory Assessment Clinic - Gainesville, Gainesville, Georgia
  - Georgia Memory Net Memory Assessment Clinic - Macon, Macon, Georgia
  - Georgia Memory Net Memory Assessment Clinic - Savannah, Savannah, Georgia
  - Georgia Memory Net Memory Assessment Clinic - Vidalia, Vidalia, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data regarding the results of longitudinal cognitive testing and functional surveys, and type, frequency, and severity of adverse events, will be available for sharing with other researchers.
Supporting Information: Study Protocol
Time Frame: Data will be made publicly available upon completion of this study and initial publication of findings from this study. Earlier access may be provided to the Centers for Medicare & Medicaid Services (CMS) or other groups who demonstrate a legitimate need for access to data.
Access Criteria: Data may be made available on request and at the discretion of the PI to CMS, other federal agencies, academic organizations, and other legitimate researchers. Data will be available for sharing for the purposes of outcome studies to evaluate the benefits and risks associated with use of lecanemab. Requests can be submitted to Georgia Memory Net (GMN) and the PI. Data request form will be made accessible on the GMN web site.
URL: https://gamemorynet.org/